CLINICAL TRIAL: NCT03288103
Title: Clinical Characterization and Trial of Growth Hormone Treatment in Patients With Aggrecan (ACAN) Deficiency
Brief Title: Growth Hormone Treatment in Patients With Aggrecan (ACAN) Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1956
Record Dates: First submitted 2017-09-18; First posted 2017-09-19 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Short Stature
MeSH Terms: conditions — Dwarfism | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Growth Hormone Treatment for Participants with ACAN Deficiency (Experimental): Pre-pubertal children with ACAN deficiency on daily growth hormone (Norditropin) regimen for a 3 year period.
  Interventions: Drug: Norditropin

INTERVENTIONS:
Drug: Norditropin — Single dose of daily growth hormone regimen. Dose will be 50 micrograms/kg/day.
  Other Names: somatropin

SUMMARY:
This is an open-label, single-arm prospective pilot study to study the effects of a single dose regimen of daily growth hormone medication (Norditropin) on pre-pubertal children with Aggrecan deficiency. The growth response will be tracked over a 12 month period. A protocol extension has been approved to continue subjects on treatment for an additional 2 years.

DETAILED DESCRIPTION:
This is a single center study. All participants will be recruited from the USA. The study intends to recruit pre-pubertal children for inclusion in the 1 year growth hormone treatment trial. The study also plans to collect the following detailed phenotypic data at the first study visit: height, weight, musculoskeletal evaluation, photographs, radiographs (knees, left hand), MRI of the knees. The participants will be required to return to Cincinnati Childrens Hospital Medical Center (CCHMC) for 3 study visits over the 12 month period. At the follow up visits participants will receive a routine physical/pubertal exam, joint exam, have vitals sign checked, height/weight taken, and labs drawn. A funduscopic exam will be performed to look for signs of intracranial pressure. Study participants are also required to complete phone check ins at scheduled intervals, and a locally drawn blood sample to check insulin-like growth factor (IGF1) levels approximately 3 months after treatment start date. Concomitant medications, adverse events will be recorded and updated at all study visits and phone check ins. Medication will be resupplied and shipped to the participant as needed at every point of follow up contact. If the subjects grow well enough in the first 12 months per study protocol, they are eligible to continue treatment through the study for an additional 2 years. They will continue to come to CCHMC every 6 months for follow up study visits. Study procedures will remain the same as the initial 1 year trial with the following additions: (1) local labs may need to be obtained for dose adjustment purposes, (2) repeat knee MRI may be completed for participants that are found to have early signs of joint disease on their baseline knee MRI scan.

The study will enroll interested and affected relatives of the participant in the joint phenotyping protocol as well. These participants will come to CCHMC only one time to complete the phenotyping visit. This is not an outcome of the study but the information gathered from the imaging will provide insight into the effects of ACAN mutation on the joint cartilage.

ELIGIBILITY:
Inclusion Criteria:

1. ACAN Deficiency - Patients must be heterozygous for a mutation in the ACAN gene. A mutation will be defined as:

   a. A heterozygous deletion of the entire gene or of >1 complete exons of the gene b. Any truncating mutation including frameshift, nonsense, splice site mutations within 2 bases of the exon/intron boundary, and start loss variants c. Any missense mutation which meets the following criteria: i. It is absent in the Exome Aggregation Consortium Database (exac.broadinstitute.org) ii. It is predicted to be damaging by both Polyphen2 and Sorting Intolerant From Tolerant (SIFT) iii. It segregates with the short stature phenotype in the family or is a de novo mutation d. In-frame insertions or deletions of >1 amino acid e. In-frame insertions or deletions of 1 amino acid must meet the same criteria as missense mutations. For the prediction programs, Alanine will be substituted for the deleted amino acid.

   f. Note - Retrospective data does not show any correlation between the type of mutation and the severity of short stature. Therefore, all mutations meeting the above criteria will be included as a single group.
2. Age - Greater than or equal to 2 years 0 days. There is no specific upper age limit, but the onset of puberty will make the patient ineligible.
3. Pre-pubertal

   1. Male subjects must have a testicular volume <4 cc as determined on physical examination by a pediatric endocrinologist at the time of the screening visit
   2. Female subjects must be Tanner 1 for breast development as determined on physical examination by a pediatric endocrinologist at the time of the screening visit
4. Bone Age - The bone age as determined by the Greulich and Pyle method must be equal to or greater than the chronological age. Bone ages will be determined at the screening visit by a single centralized radiologist.
5. Insulin-like growth factor (IGF-I) level within normal range for age and sex.
6. Ability to provide informed consent before any trial-related activities
7. Note - There is no specific height standard deviation criteria for inclusion in this study.

Exclusion Criteria:

1. Prior treatment with any of the following therapies:

   A. Growth hormone B. Insulin-like Growth Factor (IGF-I) C. Gonadotropin releasing hormone (GnRH) analog D. Aromatase Inhibitor E. Oxandrolone
2. History of any type of malignancy
3. Growth plate fusion - Defined as a bone age via the Greulich and Pyle method of 13 years in females and 15 years in males
4. Chronic medical condition known to affect growth including but not limited to:

   A. Cystic fibrosis B. Diabetes C. Inflammatory Bowel Disease D. Celiac Disease E. Asthma requiring a daily inhaled steroid dose > 400 micrograms of inhaled budesonide per day or equivalent F. Taking daily oral glucocorticoids for any reason G. Note - attention deficit hyperactivity disorder (ADHD) treated with a stimulant and treated hypothyroidism with a normal thyroid stimulating hormone (TSH) will not exclude the subject from participating in the trial.
5. (BMI) <5th percentile (CDC growth charts)
6. Any clinically significant abnormality on screening laboratory tests as determined by the principal investigator.
7. Known or suspected allergy to trial medication, excipients, or related products.
8. Contraindications to study medications, worded specifically as stated in the product's prescribing information.
9. The receipt of any investigational drug within 90 days prior to this trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Backeljauw, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Potential to share de-identified data with the primary Endocrinologist in charge of participant's clinical care

REFERENCES:
- [Result] Alexandrou E, Dauber A, Tyzinski L, Hwa V, Andrew M, Kim H, Elangovan S, Gubanich P, Taylor-Haas JA, Paterno M, Backeljauw P. Clinical phenotype and musculoskeletal characteristics of patients with aggrecan deficiency. Am J Med Genet A. 2022 Apr;188(4):1193-1203. doi: 10.1002/ajmg.a.62639. Epub 2022 Jan 9. PMID 35001504
- [Result] Muthuvel G, Dauber A, Alexandrou E, Tyzinski L, Andrew M, Hwa V, Backeljauw P. Treatment of Short Stature in Aggrecan-deficient Patients With Recombinant Human Growth Hormone: 1-Year Response. J Clin Endocrinol Metab. 2022 Apr 19;107(5):e2103-e2109. doi: 10.1210/clinem/dgab904. PMID 34922359

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total number of participants enrolled was 22, including 12 pediatric participants, and 10 adult participants. Only 10 of the pediatric patients were eligible to participate in the treatment arm of the study.
Groups:
- Treatment Group: Patients with Aggrecan (ACAN) deficiency treated with human growth hormone (rHGH) for 3 years.
- Pediatric Phenotype Group: First degree pediatric relatives of patients in the treatment group who also have Aggrecan (ACAN) deficiency but did not participate in the treatment trial.
- Adult Phenotype Group: First degree adult relatives of patients in the treatment group who also have Aggrecan (ACAN) deficiency but did not participate in the treatment trial.
Period: Overall Study
Arm/Group | Treatment Group | Pediatric Phenotype Group | Adult Phenotype Group
Started | 10 | 2 (The 12 pediatric phenotype participants includes the 10 patients in the treatment arm.) | 10
Completed | 10 | 2 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Patients with Aggrecan (ACAN) deficiency who have been treatment with human growth hormone (rHGH) for 3 years. All patients who participated in the treatment group also participated in the phenotype arm of the study.
- Phenotype Only Group: First degree relatives of patients in the treatment group who also have Aggrecan (ACAN) deficiency but did not participate in the treatment trial. Includes child and adult relatives. In total there are 22 participants in the phenotype arm, and 10 of those are also in the treatment arm.
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Phenotype Only Group | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 2 | 12
  Between 18 and 65 years | 0 | 10 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 11 | 20
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Participants in this study were recruited from across the United States
  participants
    United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Height Standard Deviation Score
Description: Height Standard Deviation Score is the standard deviation above or below the mean the height is for age and gender. Values were obtained by plotting heights on Centers for Disease Control and Prevention growth charts. An increase in Height Standard Deviation Score correlates with increase in height. Results are reported for 10 patients treated with recombinant human growth hormone.
Time Frame: Annually through three years of treatment
Population: 10 pre-pubertal children with Aggrecan deficiency
Measure: Median (Full Range); unit: standard deviation score
Groups:
- Growth Hormone Treatment for Participants With ACAN Deficiency: Pre-pubertal children with ACAN deficiency on daily growth hormone (Norditropin) regimen for a 3 year period.
  Norditropin: Single dose of daily growth hormone regimen. Dose will be 50 micrograms/kg/day, adjusted as needed per Insulin-like growth factor 1 (IGF-I) safety monitoring.
Arm/Group | Growth Hormone Treatment for Participants With ACAN Deficiency
Number analyzed (Participants) | 10
standard deviation score
  Baseline | -2.52 [-4.27 to -1.07]
  Year 1 | -1.57 [-3.89 to -0.46]
  Year 2 | -1.19 [-3.55 to -0.08]
  Year 3 | -1.09 [-3.45 to -0.02]

2. Primary Outcome: Height Velocity After Three Years of Treatment With Recombinant Human Growth Hormone (rhGH)
Description: A participants calculated height velocity derived from height measurements taken over a period of 36 months (baseline visit to 36 month visit). Only those in the treatment arm were treated with growth hormone and observed for response.
Time Frame: Annually through three years of treatment
Measure: Median (Full Range); unit: cm/year
Groups:
- Growth Hormone Treatment for Participants With ACAN Deficiency: Pre-pubertal children with ACAN deficiency on daily growth hormone (Norditropin) regimen for a 3 year period.
  Norditropin: Single dose of daily growth hormone regimen. Dose will be 50 micrograms/kg/day, adjusted if need per IGF-I safety monitoring.
Arm/Group | Growth Hormone Treatment for Participants With ACAN Deficiency
Number analyzed (Participants) | 10
cm/year
  Baseline | 5.2 [3.8 to 7.1]
  Year 1 | 8.3 [7.3 to 11.2]
  Year 2 | 7.7 [5.9 to 8.8]
  Year 3 | 6.8 [4.9 to 7.2]

3. Secondary Outcome: Number of Participants With Clinical Features of ACAN Deficiency - Osteochondritis Dissecans
Description: Evidence of osteochondritis dissecans on MRI (in those who could cooperate to perform such unsedated between the ages of 6 years-old and 20 years-old) or radiograph examination of affected participant's knees.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Pediatric Phenotype Group: This groups includes the 10 patients in the Treatment Arm and affected first degree pediatric relatives.
- Adult Phenotype Group: This include affected first degree adult relatives of the participants in the treatment arm.
Arm/Group | Pediatric Phenotype Group | Adult Phenotype Group
Number analyzed (Participants) | 12 | 10
participants | 3 | 1

4. Secondary Outcome: Number of Participants With Clinical Features of ACAN Deficiency - Osteoarthritis
Description: Evidence of early joint pathology evident (osteoarthritis) on MRI (in those who could cooperate to perform such unsedated between the ages of 6 years-old and 20 years-old) or radiograph examination of affected participant's knees, performed in those who were age appropriate and would cooperate.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Pediatric Phenotype Group | Adult Phenotype Group
Number analyzed (Participants) | 12 | 10
participants | 0 | 8

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for treatment group participants from the time of enrollment until 3 months post treatment discontinuation. Adverse event data for phenotype participants was collected from time of enrollment until one week after the completion of their one-time study visit.
Description: The definition of adverse event and/or serious adverse events does not differ from that of www.clinicialtrials.gov.
Groups:
- Treatment Group: Patients with Aggrecan (ACAN) deficiency who have been treatment with human growth hormone (rHGH) for 3 years.
- Phenotype Group: First degree relatives of patients in the treatment group who also have Aggrecan (ACAN) deficiency but did not participate in the treatment trial.
Arm/Group | Treatment Group | Phenotype Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 10/10 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=10) | Phenotype Group (N=12)
Significant behavioral changes (General disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Fever (Infections and infestations) | 3 (3) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Ear Infection (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Injection site reaction (hives) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 4 (5) | 0 (0)
Face tingling (Vascular disorders) | 1 (1) | 0 (0)
Pes planus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Injection site reaction (bruising) (General disorders) | 1 (1) | 0 (0)
Ankle Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Vomiting (General disorders) | 2 (2) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Dog bite on right ear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Root Canal (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Lipohypertrophy of upper arms (bilateral) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore Throat (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stomach pain/discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Contusion right leg (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration above left eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Medication for injection was cloudy (Product Issues) | 1 (1) | 0 (0)
Paronychia (big toe) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vaginal Yeast Infection (Infections and infestations) | 1 (1) | 0 (0)
Eyelid Erythema (Eye disorders) | 1 (1) | 0 (0)
Idiopathic Uticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Molluscum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Right Knee Injury (Abnormal ACL) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03288103/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT03288103/ICF_001.pdf